CLINICAL TRIAL: NCT05370391
Title: Comprehensive Behavioral Intervention for Tics (CBIT) for Youth With Tics and Related Emotional Disorders
Brief Title: Comprehensive Behavioral Intervention for Tics
Acronym: CBIT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Jill May Ehrenreich, Professor, Department of Psychology, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20210853
Record Dates: First submitted 2022-04-12; First posted 2022-05-11 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Tic Disorders
MeSH Terms: conditions — Tic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Comprehensive Behavioral Intervention for Tics (CBIT) (Experimental): Experimental: Comprehensive Behavioral Intervention for Tics (CBIT) Group
  Participants in this group will receive the CBIT intervention for up to 6 weeks.
  Interventions: Behavioral: Comprehensive Behavioral Intervention for Tics (CBIT)

INTERVENTIONS:
Behavioral: Comprehensive Behavioral Intervention for Tics (CBIT) — The CBIT (or CBIT-JR) intervention consists of a minimum of 6 sessions of 50-minutes each week in an individual or group setting.

SUMMARY:
The purpose of this protocol is to examine treatment outcomes of youth receiving the Comprehensive Behavioral Intervention for Tics (CBIT) and better understand the predictors, moderators, mediators and/or mechanisms of change for this intervention.

ELIGIBILITY:
Inclusion criteria

* A current diagnosis of a Diagnostic and Statistical Manual of Mental Disorders (DSM)-5 Tic disorder (e.g., Tourette's Disorder/syndrome, Persistent (Chronic) Motor or Vocal Tic Disorder, or Provisional Tic Disorder) or caregiver/youth report of clinically impairing tic symptoms
* Ability for youth to speak/read English sufficiently
* At least one parent/caregiver available to sign study consent forms, remain present during assessments, and fill out study questionnaires in English.

Exclusion criteria

* A current diagnosis of psychosis, bipolar disorder, intellectual disability, acute suicidality, alcohol/substance dependence, or eating disorder.
* Youth currently receiving psychotherapy elsewhere and/or have previously received CBIT.
* Currently suicidal or who have engaged in suicidal behaviors within the past 6 months will be excluded
* Youth currently taking psychotropic medication for a co-morbid psychiatric illness will be included without a wash-out period (to not delay treatment).

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2022-09-09 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Clinical Global Impression (CGI) - Severity Scale Scores | Change from baseline CGI-S scores to 12 weeks.
  A single-item clinician-reported measure used to assess the severity of the youth's illness at the time of assessment. The CGI-S is rated on a 7-point scale ranging from 1 (slight psychiatric illness) to 7 (extremely severe psychiatric illness). Higher scores indicate greater symptom severity.
Clinical Global Impression (CGI) - Improvement Scores | Change from baseline CGI-I scores to 12 weeks from the start of treatment.
  A single-item clinician-reported measure used to assess clinical changes in youth symptomology over the course of treatment. The CGI-I is rated on a 7-point scale ranging from 1 (very much improved since the initiation of treatment) to 7 (very much worse since the initiation of treatment). Higher scores indicate greater symptom improvement since baseline
Parent Tic Questionnaire (PTQ) | Change from pre-screen PTQ scores, to baseline, to 6 weeks, and 12 weeks from the start of treatment.
  A 28-item parent-reported measure used to assess the frequency and intensity of different motor and vocal tic symptoms in youth. The PTQ evaluates tic frequency on a 4-point scale, ranging from 1 (constant) to 4 (weekly), and intensity on a 3-point scale, ranging from 1 (mild) to 3 (very noticeable). This is done for each presenting tic. Composite total scores on the PTQ range from 2-138. Higher summed composite score indicating more tics.
Premonitory Urge Tic Scale (PUTS) | Change from baseline PUTS scores, to 6 weeks, to 12 weeks from the start of treatment.
  A 10-item self-reported measure that assess the severity of premonitory urges. The PUTS is rated on a 4-point scale ranging from 1 (not at all true) to 4 (very much true). Total scores range from 10-40 with higher scores indicating greater symptom severity.
Youth Quality of Life (YQOL) Instrument - Short Form (SF) Scores | Change from baseline YQOL Scores, to 6 weeks, to 12 weeks from the start of treatment.
  A 15-item self-reported measure of quality of life for youth ages 11-18. The YQOL-SF is rated on a 10-point scale from 0 (not at all) to 10 (very much). Scores range from 0 to 100, with higher scores indicating a higher quality of life.
Yale Global Tic Severity Scale (YGTSS) - Total Tic Scores | Change from pre-screen YGTSS Total Tic Scores, to 6 weeks, and 12 weeks from the start of treatment.
  The YGTSS is a clinician-rated interview assessing both motor and phonic tic symptoms across 5 domains: total number, frequency, intensity, complexity, and interference. Items from each domain for motor and phonic tics are summed to produce the YGTSS Total Tic Score, which ranges from 0-50. Higher scores on the YGTSS - Total Tic Score suggests greater tic severity.
Yale Global Tic Severity Scale (YGTSS) - Total Motor Tic Scores | Change from pre-screen YGTSS Total Motor Tic Scores, to 6 weeks, and 12 weeks from the start of treatment.
  The YGTSS is a clinician-rated interview assessing both motor and phonic tic symptoms across 5 domains: total number, frequency, intensity, complexity, and interference. Items from each domain for motor tics are summed to produce the YGTSS Total Motor Tic Score, which ranges from 0-25. Higher scores on the YGTSS - Total Motor Score suggests greater motor tic severity.
Yale Global Tic Severity Scale (YGTSS) - Total Phonic Tic Score | Change from pre-screen YGTSS Total Phonic Tic Scores, to 6 weeks, and 12 weeks from the start of treatment.
  The YGTSS is a clinician-rated interview assessing both motor and phonic tic symptoms across 5 domains: total number, frequency, intensity, complexity, and interference. Items from each domain for phonic tics are summed to produce the YGTSS Total Phonic Tic Score, which ranges from 0-25. Higher scores on the YGTSS - Total Phonic Score suggests greater phonic tic severity.
Yale Global Tic Severity Scale (YGTSS) - Overall Tic Related Impairment Scores | Change from YGTSS Overall Tic Related Impairment Scores pre-screen, to 6 weeks, and 12 weeks from the start of treatment.
  The YGTSS is a clinician-rated interview assessing both motor and phonic tic symptoms across 5 domains: total number, frequency, intensity, complexity, and interference. The YGTSS includes a separate impairment scale that reflects overall tic-related impairment, ranging from 0-50. Higher scores on this scale suggests greater tic impairment.
Yale Global Tic Severity Scale (YGTSS) - Global Severity Score | Change from pre-screen YGTSS Global Severity Score, to 6 weeks, and 12 weeks from the start of treatment.
  The YGTSS is a clinician-rated interview assessing both motor and phonic tic symptoms across 5 domains: total number, frequency, intensity, complexity, and interference. The YGTSS includes a separate global severity scale that ranges from 0-100. Higher scores on this scale suggests greater global tic severity.

SECONDARY OUTCOMES:
Revised Children's Anxiety and Depression Scale - Child and Revised Parent Short (RCADS-25/RCADS-P-25) Scores | Change from baseline RCADS-P scores, to 6 weeks, to 12 weeks from the start of treatment.
  A 25-item self- and parent-reported scales measuring symptoms of anxiety and depression in youth. Items are rated on a 4-point scale from 1 (Never) to 4 (always) with scores ranging from 0 to 75. A score of 70 or higher indicates high severity, above clinical threshold.
Tic Accommodation and Reactions Scale (TARS) Scores | Change from baseline TARS scores, to 6 weeks, to 12 weeks from the start of treatment.
  A 35-item parent-reported measure used to assess reactions and consequences that occur in response to youth' tics. Items focus on events at home, in school, and in other public places. The TARS is rated on a 4-point scale from 0 (not at all in the past week) to 3 (many times in the past week). Scores range from 0 to 105, with higher scores indicating greater frequency of reaction and consequences in response to their child's tics.

CONTACTS AND LOCATIONS:
Overall Officials: Jill Ehrenreich-May, Ph.D., Study Director — University of Miami
Locations (1):
- University of Miami, Coral Gables, Florida, United States

IPD SHARING:
Plan to Share IPD: No